CLINICAL TRIAL: NCT06740773
Title: A Retrospective Study to Identify Risk Factors for Complications After Cranioplasty
Brief Title: Risk Factors for Complications After Cranioplasty
Status: Recruiting | Type: Observational
Sponsor: Qilu Hospital of Shandong University (Other)
Collaborators: Daping Hospital of Army Medical University (Other); Tang-Du Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KYLL-202407-041
Record Dates: First submitted 2024-12-11; First posted 2024-12-18 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2024-12

CONDITIONS: Cranioplasty; Postoperative Complications; Risk Assessment
Keywords: Cranioplasty; Postoperative Complications; Risk factors; Retrospective Study; predictive model
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Derivation Cohort: Identification of risk factors, development and internal validation of predictive models
- External Validation Cohort: External validation of the predictive models

SUMMARY:
Cranial defects often result from brain injuries, hemorrhages, strokes, or brain tumors. These conditions can increase pressure inside the skull, and if left untreated, may lead to dangerous complications like brain herniation. To manage this, a common procedure called decompressive craniectomy is performed to reduce intracranial pressure. While this surgery often stabilizes the patient's condition, it leaves a cranial defect that exposes the brain to external risks, including pressure fluctuations and potential damage. In severe cases, patients with larger defects may develop complications such as sinking skin flap syndrome.

Cranial reconstruction, also known as cranioplasty, is an important procedure to restore the skull's structure and protect the brain. This surgery can improve brain function, stabilize intracranial pressure, and enhance the patient's appearance. While cranioplasty is a standard neurosurgical procedure, it has a relatively high risk of complications compared to other brain surgeries. Common complications include infections, bleeding, hydrocephalus, and seizures. In severe cases, complications may lead to the failure of the reconstruction.

Understanding the factors that contribute to complications after cranioplasty is crucial for neurosurgeons to improve outcomes and reduce risks. This study aims to identify these factors and develop predictive models for postoperative complications of cranioplasty.

DETAILED DESCRIPTION:
Cranial defects, often caused by conditions such as traumatic brain injuries, strokes, or brain tumors, present a significant clinical challenge. Decompressive craniectomy, frequently performed to manage increased intracranial pressure, leaves patients with cranial defects that require subsequent cranioplasty. Cranioplasty, while being a common neurosurgical procedure, has a higher complication rate compared to other cranial surgeries, warranting a deeper investigation into its risk factors.

In addition to identifying risk factors, this study aims to develop and validate predictive models for postoperative complications. Advanced statistical techniques, such as machine learning algorithms, will be used to assess the contribution of individual variables to complication risk.

By leveraging a large multi-center dataset, the study seeks to provide actionable insights into the prevention of postoperative complications. The results are expected to inform clinical decision-making, enhance patient outcomes, and improve the quality of perioperative care in neurosurgical practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent cranioplasty in the Department of Neurosurgery at Qilu Hospital of Shandong University, Tangdu Hospital of Air Force Medical University, or Daping Hospital, Army Military Medical University between January 1, 2015, and July 31, 2023
* Diagnosed with cranial defects
* Possessed complete and accessible electronic medical records
* Patients had no prior history of cranioplasty

Exclusion Criteria:

* Patients with a prior history of cranioplasty
* Severe comorbidities (such as serious cardiac, liver, kidney and immune system dysfunction)
* Congenital cranial defects
* Severe missing data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with cranial defects who underwent their first cranioplasty in the Department of Neurosurgery at Qilu Hospital of Shandong University between January 1, 2015, and January 1, 2025, or at Tangdu Hospital of Air Force Medical University or Daping Hospital of the Army Medical University between January 1, 2015, and July 31, 2023.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Risk factors for postoperative complications of cranioplasty | From the date of cranioplasty to the date of hospital discharge, with complications assessed throughout the hospitalization period, up to 60 days.
  The primary outcome is to identify factors associated with postoperative complications of cranioplasty. The analysis will focus on patient demographics, comorbidities, surgical details, and other clinical variables extracted from medical records

SECONDARY OUTCOMES:
Establishment predictive models for postoperative complications of cranioplasty | From the date of cranioplasty to the date of hospital discharge, with complications assessed throughout the hospitalization period, up to 60 days.
  The secondary outcome is to develop and validate predictive models for postoperative complications of cranioplasty based on identified risk factors.

CONTACTS AND LOCATIONS:
Overall Officials: Ning Yang, M.D., Ph.D, Principal Investigator — Department of Neurosurgery, Qilu Hospital of Shandong University
Locations (3):
- China (3):
  - Department of Neurosurgery, Daping Hospital of Army Medical University, Chongqing, Chongqing Municipality
  - Department of Neurosurgery, Tang-Du Hospital, Xi'an, Shaanxi
  - Department of Neurosurgery, Qilu Hospital of Shandong University, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD
Supporting Information: Study Protocol, Analytic Code
Time Frame: Beginning 1 year after publication with no end date
Access Criteria: The individual participant data (IPD) and supporting information are available from the corresponding author upon reasonable request via email. Access will be provided to researchers with a scientifically sound proposal and for non-commercial purposes, in compliance with ethical guidelines.

REFERENCES:
- [Result] Bader ER, Kobets AJ, Ammar A, Goodrich JT. Factors predicting complications following cranioplasty. J Craniomaxillofac Surg. 2022 Feb;50(2):134-139. doi: 10.1016/j.jcms.2021.08.001. Epub 2021 Aug 25. PMID 34580005
- [Result] Chaturvedi J, Botta R, Prabhuraj AR, Shukla D, Bhat DI, Devi BI. Complications of cranioplasty after decompressive craniectomy for traumatic brain injury. Br J Neurosurg. 2016;30(2):264-8. doi: 10.3109/02688697.2015.1054356. Epub 2015 Jun 17. PMID 26083136
- [Result] Zanaty M, Chalouhi N, Starke RM, Clark SW, Bovenzi CD, Saigh M, Schwartz E, Kunkel ES, Efthimiadis-Budike AS, Jabbour P, Dalyai R, Rosenwasser RH, Tjoumakaris SI. Complications following cranioplasty: incidence and predictors in 348 cases. J Neurosurg. 2015 Jul;123(1):182-8. doi: 10.3171/2014.9.JNS14405. Epub 2015 Mar 13. PMID 25768830
- [Result] Belzberg M, Mitchell KA, Ben-Shalom N, Asemota AO, Wolff AY, Santiago GF, Shay T, Huang J, Manson PN, Brem H, Gordon CR. Cranioplasty Outcomes From 500 Consecutive Neuroplastic Surgery Patients. J Craniofac Surg. 2022 Sep 1;33(6):1648-1654. doi: 10.1097/SCS.0000000000008546. Epub 2022 Mar 4. PMID 35245275
- [Result] Malcolm JG, Rindler RS, Chu JK, Grossberg JA, Pradilla G, Ahmad FU. Complications following cranioplasty and relationship to timing: A systematic review and meta-analysis. J Clin Neurosci. 2016 Nov;33:39-51. doi: 10.1016/j.jocn.2016.04.017. Epub 2016 Aug 4. PMID 27499122
- [Result] Singh S, Singh R, Jain K, Walia B. Cranioplasty following decompressive craniectomy - Analysis of complication rates and neurological outcomes: A single center study. Surg Neurol Int. 2019 Jul 19;10:142. doi: 10.25259/SNI_29_2019. eCollection 2019. PMID 31528477
- [Result] Honeybul S, Ho KM. Long-term complications of decompressive craniectomy for head injury. J Neurotrauma. 2011 Jun;28(6):929-35. doi: 10.1089/neu.2010.1612. Epub 2011 Jun 1. PMID 21091342
- [Result] Henry J, Amoo M, Murphy A, O'Brien DP. Complications of cranioplasty following decompressive craniectomy for traumatic brain injury: systematic review and meta-analysis. Acta Neurochir (Wien). 2021 May;163(5):1423-1435. doi: 10.1007/s00701-021-04809-z. Epub 2021 Mar 23. PMID 33759012